CLINICAL TRIAL: NCT00308880
Title: If Tranexamic Acid Could Reduce the Duration of Drainage Tube Placement ? -A Prospective Randomized Study in Head and Neck Surgery Patients
Brief Title: Tranexamic Acid and Head and Neck Surgery Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCVGH-957001A; 941117/C05186
Record Dates: First submitted 2006-03-29; First posted 2006-03-30 (Estimated); Last update posted 2006-03-30 (Estimated); Status verified 2006-03

CONDITIONS: Head and Neck Neoplasms
Keywords: Tranexamic acid; head neck surgery
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Tranexamic Acid

INTERVENTIONS:
Drug: Transamin

SUMMARY:
Tranexamic acid belongs to fibrinolytic inhibitors. Several prospective randomized clinical trials have proved its effectiveness in reducing intra-operative and post-operative bleeding in orthopedic and cardiovascular surgeries. However, there is little study about tranexamic acid in reducing post-operative bleeding in head and neck surgery. So the aim of this study is to investigate if tranexamic acid could reduce post-operative bleeding via prospective double-blinded randomized clinic trial.

DETAILED DESCRIPTION:
Otolaryngologists often use drainage tube after head and neck surgery to reduce hematoma or seroma formation. In addition, the duration of drainage tube placement is closely related to the length of hospital stay. So early removal of drainage tube could eventually shorten the admission period. The factors related to the duration of drainage tube placement include: type of surgery, intra-operative bleeding, underlying disease of coagulation disorders, etc. According to the literatures, the average duration of drainage in head and neck surgery is 4 days. Another study showed that one of the risk factors associated with surgical site infection is the longer drainage duration. Therefore, how to remove drainage tube as soon as possible is crucial to head and neck surgeon.Tranexamic acid belongs to fibrinolytic inhibitors. Several prospective randomized clinical trials have proved its effectiveness in reducing intra-operative and post-operative bleeding in orthopedic and cardiovascular surgeries. However, there is little study about tranexamic acid in reducing post-operative bleeding in head and neck surgery. So the aim of this study is to investigate if tranexamic acid could reduce post-operative bleeding via prospective double-blinded randomized clinic trial.This study includes 60 consecutive patients who will undergo head and neck surgery. Those who are allergy to tranexamic acid, history of coagulation disorders, under anti-coagulation therapy will be excluded. Basic data will be recorded along with detail physical examination and operation type. Then they will be divided randomly into study group and control group. Study group will receive tranexamic acid before and after operation while control group not. PT, APTT, level of prothrombin fragments 1+2, D-dimers, plasminogen, α2-antiplasmin, tissue plasminogen activator (tPA), and plasminogen activator inhibitor (PAI-1) will be obtained before and after operation. The drainage amount, duration of drainage tube placement will also be recorded. Relevant variables will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* head and neck neoplasm scheduled for operation

Exclusion Criteria:

* allergy to tranexamic acid
* history of coagulation disorders
* under anti-coagulation therapy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2006-03; Study Completion 2007-03

PRIMARY OUTCOMES:
Drainage amount
Drainage stay duration
Laboratoy data

CONTACTS AND LOCATIONS:
Overall Officials: Shih-An Liu, MD, MHA, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan